CLINICAL TRIAL: NCT01527370
Title: A Phase III Clinical Trial to Study the Safety, Tolerability, and Immunogenicity of ZOSTAVAX™ in Healthy Adults in India
Brief Title: Safety, Tolerability, and Immunogenicity of Zoster Vaccine Live (ZOSTAVAX™) in Healthy Adults in India (V211-025)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V211-025; CTRI/2012/08/002922 (Registry Identifier: CTRI)
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Herpes Zoster; Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zoster Vaccine Live (Experimental)
  Interventions: Biological: Zoster Vaccine Live

INTERVENTIONS:
Biological: Zoster Vaccine Live — One approximately 0.65 mL injection subcutaneously on Day 1
  Other Names: ZOSTAVAX™; V211

SUMMARY:
This study will determine if ZOSTAVAX™ is safe, tolerable, and immunogenic in healthy adults in India.

ELIGIBILITY:
Inclusion Criteria:

* No fever on day of vaccination
* Females have a negative pregnancy test and use an acceptable method of birth control, or are postmenopausal
* Underlying chronic illnesses must be stable

Exclusion Criteria:

* History of hypersensitivity reaction to any vaccine component
* Prior receipt of a varicella or zoster vaccine
* Prior history of herpes zoster
* Have recently had another vaccination
* Have recently received blood products other than autologous blood transfusion
* Pregnant or breast feeding
* Use of immunosuppressive therapy
* Known or suspected immune dysfunction
* Use of nontopical antiviral therapy with activity against herpesvirus

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2013-04-09 (Actual); Study Completion 2013-04-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sreenivasamurthy L, Pandey S, Chandra BS, Sharma M, Ranganathaiah SR, Vaidya P, Naik R. Immunogenicity, Safety, and Tolerability of Live Attenuated VaricellaZoster Virus Vaccine (ZOSTAVAX) in Healthy Adults in India. J Assoc Physicians India. 2018 Jul;66(7):50-54. PMID 31325263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten sites in India enrolled adult participants in the study.
Groups:
- Zoster Vaccine Live: A single dose of Zoster vaccine was administered on day 1. Participants were followed up to day 42 for safety and immunogenicity.
Period: Overall Study
Arm/Group | Zoster Vaccine Live
Started | 250
Completed | 244
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 184

OUTCOME MEASURES:

1. Primary Outcome: The Geometric Mean Titer (GMT) of Varicella-zoster Virus (VZV) Antibody at 6 Weeks Postvaccination
Description: Antibody titers were measured by VZV-specific glycoprotein enzyme-linked immunosorbent assay (gpELISA).
Time Frame: Prevaccination up to 6 weeks postvaccination
Population: This endpoint was analyzed in the per-protocol population which included all participants who were vaccinated and had no major deviations from the protocol procedure. At the week 6 postvaccination timepoint, a total of 7 participants were excluded from the per-protocol immunogenicity analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 250
gpELISA units/mL
  Prevaccination (n=250) | 149.8 [132.6 to 169.2]
  6 weeks postvaccination (n=243) | 410.8 [373.0 to 452.6]

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titers at 6 Weeks Postvaccination
Description: GMFR was analyzed as the geometric mean of the ratio of VZV antibody titer (gpELISA units/mL) at postvaccination week 6 over VZV antibody titer (gpELISA units/mL) at prevaccination day 1.
Time Frame: Prevaccination up to 6 weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 243
Ratio | 2.8 [2.5 to 3.1]

3. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event is one that results in death, is life-threatening, results in a persistent or significant disability, results in or prolongs hospitalization, results in a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgment.
Time Frame: Up to 42 days postvaccination
Population: This endpoint was analyzed in all participants who were vaccinated and had any safety follow up data.
Measure: Number; unit: Participants
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 250
Participants | 2

ADVERSE EVENTS:
Time Frame: Day 1 up to day 42 postvaccinaton
Description: Adverse events were collected from all participants who were vaccinated and had any safety follow up data.
Arm/Group | Zoster Vaccine Live
Serious Adverse Events (participants affected / at risk) | 2/250
Other Adverse Events (participants affected / at risk) | 47/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster Vaccine Live (N=250)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster Vaccine Live (N=250)
Injection site erythema (General disorders) | 35 (36)
Injection site pain (General disorders) | 22 (24)
Injection site swelling (General disorders) | 31 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.